CLINICAL TRIAL: NCT05150366
Title: Impact of Percutaneous Closure of the Left Atrial on the Maximum Proto-diastolic Speed of the Mitral Ring Measured by Tissue Doppler
Brief Title: Impact of Percutaneous Closure of the Left Atrial on the Maximum Proto-diastolic Speed of the Mitral Ring Measured by Tissue Doppler (ACTIFER)
Acronym: ACTIFER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-A02663-36
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Tissue Doppler; Left Atrial Closure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient scheduled for percutaneous closure of the left auricle by St Jude AMULET device (Experimental)
  Interventions: Procedure: Trans thoracic echocardiography

INTERVENTIONS:
Procedure: Trans thoracic echocardiography — trans thoracic echocardiography at the beggining and at the end of the placement of the Saint Jude Medical AMULET type prosthesis

SUMMARY:
The main objective is to demonstrate the equivalence, before and after the percutaneous closure of the left atrial procedure, of the maximum proto-diastolic velocity of the lateral mitral annulus (e 'lat) measured by tissue Doppler. Patients with AF at high embolic risk and presenting a formal and definitive contraindication to anticoagulants having been operated on for percutaneous closure of the left atrial by St Jude AMULET device, considering an equivalence margin of 1 cm / sec.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years-old
* Patient with paroxysmal AF at high embolic risk (CHA2DS2Vasc score ≥ 4) and presenting a formal and definitive contraindication to anticoagulants
* Patient scheduled for percutaneous closure of the left auricle by St Jude AMULET device
* Patient in sinus rhythm
* Subject affiliated or beneficiary of a social security scheme
* Patient having signed the informed consent

Exclusion Criteria:

* Patient participating in another clinical study
* Patient in permanent ACFA
* Patient with a mitral prosthesis (biological or mechanical),
* Patient with a history of mitral annuloplasty
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision;
* Pregnant, breastfeeding or parturient woman;
* Patient hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-09-17 (Estimated); Study Completion 2022-09-17 (Estimated)

PRIMARY OUTCOMES:
lateral e' speed | 1 day
  measured by tissue Doppler

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Le Bois, Lille, France